CLINICAL TRIAL: NCT06746623
Title: Nonendoscopic Screening for Barrett's Esophagus and Esophageal Cancer in At-Risk Veterans Without History of Chronic Gastroesophageal Reflux
Brief Title: Nonendoscopic Screening for Barrett's Esophagus in Veterans Without Chronic Reflux
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Louis Stokes VA Medical Center (U.S. Federal Agency)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Katarina Greer, Gastroenterologist, Associate Professor of Medicine, Louis Stokes VA Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DOD HT94252410741
Record Dates: First submitted 2024-11-15; First posted 2024-12-24 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-04

CONDITIONS: Obese Patients; Tobacco Use; Veterans; Family History of Esophageal Cancer; Barrett Esophagus
Keywords: Non-endoscopic screening; esophagus; Barrett
MeSH Terms: conditions — Tobacco Use; Barrett Esophagus

STUDY DESIGN:
Masking Description: Participants will complete screening for the condition by completing bedside Esocheck test and upper endoscopy. Providers performing endoscopy will not have result of Esocheck test available to them when performing upper endoscopy. Lab analysis team will not have endoscopy and histology results available to them to interpret methylation status results or Esoguard assay.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- This is a single arm study. Participants will complete 2 diagnostic tests: Esocheck and EGD. (Other): Patients without history of GERD receiving care in Wade Park VA will be approached regarding BE screening. Reasons for refusal of screening will be recorded. Adult subjects without history of gastroesophageal reflux with three or more risk factors- white race, male gender, obesity (BMI > 30), smoking, or family history will be included. Only those patients who have not had prior EGD will be candidates for Esocheck screening. Distal esophageal samples will be assayed for mVIM + mCCNA1 (Esoguard assay). All patients will be offered upper endoscopy.
  Interventions: Diagnostic Test: Enrolled participants will complete Esocheck/Esoguard and diagnostic upper endoscopy.

INTERVENTIONS:
Diagnostic Test: Enrolled participants will complete Esocheck/Esoguard and diagnostic upper endoscopy. — Esocheck (EC)/Esoguard (EG): EC is a encapsulated balloon device available commercially from Lucid Diagnostics (New York, NY). EG assay uses bisulfite sequencing for detection of aberrant methylation in the vimentin and cyclin A1 genomic loci, respectively.
  EGD (upper endoscopy): EGD will be performed by gastroenterologists practicing in the Louis Stokes Cleveland VA Medical Center Endoscopy laboratories on the same day when EC/EG is performed.

SUMMARY:
The veteran population is at increased risk for EAC and its precursor lesion, Barrett's esophagus (BE), due to increased prevalence of disease risk factors compared to the general population. BE is traditionally diagnosed only when patients undergo endoscopy with biopsies. However, due to the high cost of endoscopy and the lack of studies proving efficacy of screening, endoscopy to screen for BE is not routinely recommended. A simpler screening procedure similar to a pap smear would be an ideal way to sample the esophageal tissue for cancer and its precursor condition, BE. This study proposes a non-endoscopic detection method administered in outpatient offices which would increase subsequent endoscopic detection of BE. The study team will be enrolling veterans who do not have history of gastroesophageal reflux but have multiple risk factors for esophageal adenocarcinoma.

DETAILED DESCRIPTION:
This research study addresses early detection of esophageal adenocarcinoma (EAC). Incidence of EAC has increased more than 6-fold in the past four decades yet prognosis for patients with EAC remains poor with less than 20% of patients surviving beyond 5 years. The veteran population is at increased risk for EAC and its precursor lesion, Barrett's esophagus (BE), due to increased prevalence of disease risk factors (age, male, obesity, smoking, family history of BE or EAC), compared to the general population. Current society guidelines recommend one-time upper endoscopy for persons with gastro-esophageal reflux (GERD) plus additional risk factors for BE and EAC. Still, up to 40% of patients who develop esophageal cancer do not report history of GERD preceding cancer diagnosis. Screening benefit needs to be explored in these patients without history of GERD.

Hypothesis: The incorporation of a non-endoscopic detection method in clinical practice will increase the positive predictive value of esophagogastroduodenoscopy (EGD) and increase the detection of BE among veterans who do not report GERD but have multiple risk factors for EAC.

Objectives: Unsedated non-endoscopic BE screening method will be offered to veterans at risk of EAC but without GERD history.

The Specific Aims are: 1. To detect BE in high-risk subjects without GERD, using a non-endoscopic biomarker-based screening tool. 2. Measure screening acceptance rate, reasons for refusal and screening yield.

Preliminary Data: Prospectively collected data from Cleveland VA showed that the sensitivity of this non-endoscopic screening tool in patients with chronic GERD and/or PPI use was 92.9% (95% CI 66.1-99.8), and specificity of 72.2% (95% CI 62.1-80.8). A retrospective study of 113 patients with EAC at Louis Stokes Cleveland VA Medical Center found that 52 (46%) presented with Stage IV disease. Of these patients with metastatic cancer who were eligible for screening, 20 (39%) had been seen in clinic at least one year prior to cancer diagnosis and had not been screened with EGD. In the overall group, 42 of the 117 patients had been seen in clinic with GERD previously and 26 (62%) had not been screened.

Research Design: Patients without history of GERD will be approached regarding BE screening. Reasons for refusal of screening will be recorded. Adult subjects without history of gastroesophageal reflux with three or more risk factors- white race, male gender, obesity (BMI > 30), smoking, or family history will be included. Only those patients who have not had prior EGD will be candidates for Esocheck screening. Distal esophageal samples will be assayed for mVIM + mCCNA1 (Esoguard assay). All patients will be asked to complete upper endoscopy.

Sample Size and Analysis: The prevalence of BE found on EGD performed in Caucasian men without chronic GERD is around 8.5%. Assuming prevalence of BE of 9%, and sensitivity/specificity of Esocheck/Esoguard equal to 90/90%, respectively, this study plans to recruit 400 patients. Sensitivity, specificity, diagnostic accuracy of Esocheck/Esoguard in patients without GERD will be calculated. Acceptance rates of screening will be reported. Latent class analysis will be performed to examine common patterns among patients who decline EAC screening.

ELIGIBILITY:
Inclusion Criteria:

* Patients without history of chronic GERD who meet criteria for upper endoscopic screening for BE will be accrued35.

  1. Adults > 40 and < 85 years old who have no prior EGD and can provide informed consent
  2. Absence of chronic GERD symptoms (absence of weekly heartburn or regurgitation, not on medications for GERD), and are:

     a. Meet ACG/AGA Clinical Guideline criteria for BE screening. Eligible subjects will have at least three additional risk factors for BE (white race, obesity defined as BMI > 30, male gender, current smoker or smoking history > 10 pack years, family history of Barrett's esophagus or EAC central obesity (waist size > 35 inches for women and > 40 inches for men), white race, male sex, confirmed history of BE/EAC in at least two family members, with one a first degree relative).
  3. No known coagulopathy, no known esophageal varices, not on chronic anticoagulation therapy, and have:
  4. No significant dysphagia or odynophagia

Exclusion Criteria:

* Exclusion Criteria

  1. History of prior EGD procedure in past ten years
  2. Inability to provide written informed consent
  3. History of weekly or more frequent heartburn or regurgitation for five or more years
  4. On anti-coagulant drug(s) that cannot be temporarily discontinued or coagulopathy with INR > 1.5
  5. Known history of esophageal varices or esophageal stricture
  6. Any contraindication, as deemed in Investigator's medical judgment, to undergoing the EsoCheck procedure, undergoing the EGD procedure, and/or having biopsies taken, including but not limited to due to comorbidities such as coagulopathy or a known history of esophageal diverticula, esophageal fistula and/or esophageal ulceration
  7. History of difficulty swallowing (dysphagia) or painful swallowing (odynophagia), including swallowing pills
  8. Oropharyngeal tumor
  9. History of esophageal or gastric surgery, with exception on uncomplicated recent surgical fundoplication procedure with documented normal acid exposure time (AET) percent (AET <4%)
  10. History of myocardial infarction or cerebrovascular accident within past 6 months

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-04-11 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Esoguard assay and histology confirming diagnosis of Barrett's esophagus and/or esophageal adenocarcinoma | Laboratory and pathology results will be finalized within 10 and up to 30 days
  Results from enrollment visit

CONTACTS AND LOCATIONS:
Overall Officials: Katarina B Greer, MD/MS, Principal Investigator — Cleveland VA Research and Education Foundation
Locations (1):
- VA Northeast Ohio Healthcare System, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Study protocol, statistical analysis plan and informed consent will be made available upon request from principal investigator. Study report will be available at the end of study period, i.e. in September of 2027.

REFERENCES:
- [Background] Greer KB, Blum AE, Faulx AL, Deming EM, Hricik LL, Siddiqui H, Wilson BM, Chak A. Nonendoscopic Screening for Barrett's Esophagus and Esophageal Adenocarcinoma in At-Risk Veterans. Am J Gastroenterol. 2025 Mar 1;120(3):545-553. doi: 10.14309/ajg.0000000000002962. Epub 2024 Jul 11. PMID 38989889